CLINICAL TRIAL: NCT05749419
Title: Questionnaires and Focus Groups Based Quantitative & Qualitative Study of Vaccine Hesitancy and Confidence Among At-risk and Marginalized Populations: Persons With Special Needs, Intellectual Disabilities and Congenital Anomalies
Brief Title: Vaccinations and People With Disabilities
Status: Recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Tenenbaum Ariel, Principal investigator, MD, Clinical Professor, Director of the center for children with chronic diseases, Hadassah Medical Organization
Other Study IDs: Tenenbaum-HMO-CTIL
Record Dates: First submitted 2023-02-08; First posted 2023-03-01 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-09

CONDITIONS: Vaccine Refusal; Compliance, Patient; Disability, Intellectual; Congenital Disorders; Pediatric Disorder
MeSH Terms: conditions — Vaccination Refusal; Patient Compliance; Intellectual Disability; Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group and control group: Study group - children with chronic diseases, disabilities, or congenital anomalies.
  Control group - their siblings.

SUMMARY:
The goal of this observational study is to learn about vaccinations hesitancy, delay or avoidance in children with chronic diseases, congenital anomalies or disabilities. The main questions it aims to answer are:

• Attitudes of caregivers towards vaccinating their children, obstacles that postpone vaccinations, and the status of vaccinations of these children.

Participants will fill out questionnaires and some will be included in focused groups for the qualitative part of the study.

Researchers will compare the vaccinations status of the research group to their siblings' status as well as the published national records of vaccination compliance.

DETAILED DESCRIPTION:
Global vaccines programs prevent infectious diseases, congenital anomalies and cancer [1,2]. Full and partial avoidance of vaccines, or postponing vaccines, may lead to morbidity, disability and mortality. This is particularly significant among children and adults with special needs, intellectual and developmental disabilities, and congenital anomalies, which are at-risk groups, together representing over 15% of the general population [3,4]. Studies have shown that this population is particularly vulnerable when it comes to infectious diseases, hospitalizations, sexually transmitted diseases, abuse and neglect [5,6,7]. Furthermore, this is a marginalized population, with (in average) a lower socioeconomic status and at a lower level of education of themselves and their caregivers [8]. The reasons for hesitance, avoidance or selectivity of vaccines by the caregivers are not comprehensively characterized. Therefore, the investigators outline our thoughts and Insights from our ongoing work, for over two decades, with this population. In the investigators experience, when doctors and nurses ask the patients and their caregivers what are the reasons for less-then-optimal vaccination state, there are several explanations: concurrent illnesses that made them postpone vaccinations, access challenges, being preoccupied with many other health tasks, and paradoxically the fear that the child is too fragile for receiving the vaccine or that the vaccine itself will do harm. Also, some may be wrongly advised about contraindications that are misinterpreted. It is surprising that the infestigators hear from caregivers about the fear from the vaccines, and not about the fear from the diseases. Another important issue is the unfortunate vulnerability of this population to STD's, which the investigators repeatedly hear from caregivers that this is a non-issue for them, which is clearly a dangerous misconception [9].

Therefore, healthcare professionals are missing valuable information about possible risks and intervention opportunities among an at-risk population.

Objectives:

1. The investigators will systematically map the reasons for the delay and/or avoidance, and/or hesitance to vaccinate by conducting a large-scale evaluation of current and planned immunizations among persons of all ages who have special needs, intellectual and developmental disabilities and congenital anomalies (study group). The investigatorswill use a comprehensive questionnaire to collect this information, as well as focused discussion groups for in-depth qualitative investigations. The investigators will compare the data with their sibling's vaccination status and with recruits from the general population (control group).

According to the concept "Do not talk about us without us", The investigators will include persons with special needs and disabilities in the study and make all efforts to hear directly from them in focus groups or individually about their approach to vaccinations, including hesitancies and misconceptions about the procedure.

Hypotheses:

1. There is a higher prevalence of vaccine avoidance and delay among the study population.
2. The reasons for avoidance and/or delay are:

A. Fear of harm - The study population are perceived more fragile, hence more likely to adversely react to vaccines.

B. Misconceptions about their vulnerability to STD's, and false beliefs about neurodevelopmental effects of the vaccines themselves.

This is a descriptive qualitative and quantitative study. The Quantitative part consists of comprehensive questionnaires that The investigators will design for the study. The questionnaire will have five sections: 1. Sociodemographic data. 2. Current vaccination status. 3. Delay/hesitancy/avoidance - past present and future plans. 4. Reasons for delay/hesitancy/avoidance if exist. 5. Statements regarding vaccines benefits, safety, known side effects, and misconceptions, and the participants' level of agreement with these statements. All questionnaires will be filled out anonymously after consent to participate.

For the focused groups The investigators will recruit parents and other caregivers as well as persons with disabilities. The investigators will analyze these opened and free discussions, with limited opening remarks and follow up questions for clarification, in a qualitative manner and all themes, dilemmas and experiences will be presented accordingly.

It is based on questionnaires and focus groups studies, with control groups. The investigators will conduct the research in the Hadassah- Hebrew university medical center, in collaboration with associations and institutions that provide healthcare and support for the studied population and their families.

Since The investigators have ongoing collaborations with other academic and clinical institutions in other countries, it is possible for us to explore with them a fruitful collaboration in this research, and developing it to a multicenter study.

The investigators hopefully plan to recruit a total of one thousand participants.

The study population is our patients and their families that arrive for evaluations and treatments. The investigators plan to recruit more participants with the collaboration other associations and institutions. The population is consisted of persons with a variety of disabilities, namely intellectual and developmental disability, Down syndrome, congenital syndromes and genetic disorders.

The investigators will try to include as many persons as possible, excluding those who are reluctant to participate or did not provide minimal information in the questionnaires.

As part of the study procedure and presentation of the results, The investigators will aim to conceptualize tailored programs to increase vaccination confidence and adherence, and propose a follow-up interventional study.

ELIGIBILITY:
Inclusion Criteria:

• Diagnosed children with disabilities, chronic diseases or congenital anomalies

Exclusion Criteria:

* Undiagnosed children
* Inadequate filled out questionnaires

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children with disabilities, chronic conditions and congenital anomalies. The parents will fiil out the questionnaires and participate in focus groups.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Percentages of children in the study group who are not vaccinated, partially vaccinated, or vaccinated late, in comparison with the percentages in the control group. | 2 years
  Percecntages as described above as well as description of reasons for vaccination avoidance, delay and hesitancy, obstacles in the way to vaccinate, approach to vaccines as detaled in the questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Tenenbaum, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah medical center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No